CLINICAL TRIAL: NCT04034732
Title: The Feasibility and Effects of Mindfulness Based Relapse Prevention (MBRP) on Reducing Craving and Addictive Behaviour in Adults With Substance Abuse Disorders
Brief Title: MBRP on Reducing Craving and Addictive Behaviour in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Daisy Dexing Zhang, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MBRP protocol version 2
Record Dates: First submitted 2019-07-18; First posted 2019-07-26 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Substance Abuse; Substance Use Disorders
Keywords: Mindfulness-based intervention; Mindfulness; Relapse prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Masking Description: In this open-label study, blinding of therapists and participants will not be possible. However, all data collection will be performed by a trained research assistant blinded to the allocation status of the participants. The research assistant will receive rigorous training in standardized data collection procedures. Data entry will be prepared so that the person can conduct the statistical analyses without referring to allocation information, thus ensuring blinding during data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Relapses Prevention (MBRP) (Experimental): The MBRP program will be delivered by an instructor with training in MBSR/MBCT who has more than two years of teaching experience in MBSR/MBCT. The MBRP programme will consist of 2.5 hour weekly sessions for 8 weeks. The mindfulness curriculum will include training in mindfulness through (1) a body scan, (2) sitting meditation and (3) mindful stretching exercises.
  Interventions: Behavioral: Mindfulness-based Relapses Prevention (MBRP)
- Usual Care Control Group (UCCG) (Active Comparator): Participants in the UCCG condition will remain in their standard outpatient aftercare provided by the treatment agency with an aim to maintain their abstinence with the help from social workers or other healthcare professionals through different activities, such as topics on life training skills such as rational thinking skills, grief and loss, assertiveness, self esteem, goal setting, effects of drugs on interpersonal relationships and experience. Frequency of their visits to / contacts with healthcare professionals will be recorded.
  Interventions: Behavioral: Usual Care Control

INTERVENTIONS:
Behavioral: Mindfulness-based Relapses Prevention (MBRP) — Manualized MBRP program is used with a central theme in each session, with meditation practices and relapse prevention exercises and discussions. Themes include the concept of "automatic pilot" and its relationship to addiction relapse, recognizing thoughts and emotions in relation to triggers of relapse, integrating mindfulness practices into daily activities, practicing mindfulness in high risk situations and the role of thoughts and emotions in relapse. Include daily homework exercises that consist of awareness exercises directed at increasing non-judgmental awareness of bodily sensations, thoughts and feelings, together with exercises designed to integrate awareness skills into daily life. Include training in mindfulness through body scan, sitting meditation, and mindful stretching exercises, to cultivate awareness during simple stretching movement.
  Arms: Mindfulness-based Relapses Prevention (MBRP)
Behavioral: Usual Care Control — Participants in the UCCG condition will remain in their standard outpatient aftercare provided by the treatment agency with an aim to maintain their abstinence with the help from social workers or other healthcare professionals through different activities, such as topics on life training skills such as rational thinking skills, grief and loss, assertiveness, self esteem, goal setting, effects of drugs on interpersonal relationships and experience. Frequency of their visits to / contacts with healthcare professionals will be recorded.
  Arms: Usual Care Control Group (UCCG)

SUMMARY:
Mindfulness-base interventions are promising interventions as an adjunctive therapy to be integrated into current existing anti-drug services. The advantages of MBRP can include: 1) having very low stigma as mindfulness courses are already widely accepted and used among different populations including healthy populations. The running of mindfulness courses can be more acceptable by the community; 2) it could be more accessible and cost-effective as it can be provided in group and in community settings; 3) it is a skill that can be learned and be used after the 8 week course , e.g. when the drug user is triggered in unforeseen circumstances, they may apply the learnt mindfulness skills to help themselves overcome the difficulties when timely professional help is not available; 4) Drug Abuse Statistics from Narcotics Division, Security Bureau of the government of Hong Kong showed that the most common reasons for recurrent drug use were to avoid discomfort of its absence (62%) and relief of depression/stress/boredom (30%).

The study objectives are as follow:

1. To evaluate the feasibility of using mindfulness- based relapse prevention (MBRP) programme among adults with substance abuse in Hong Kong;
2. To examine the changes of craving, substance use, mood symptoms, self-efficacy, acceptance, level of mindfulness and quality of life between those who have enrolled in the MBRP as compared to those in the usual care control group;
3. To evaluate the correlations between changes in substance use and craving and changes in mood symptoms, self-efficacy, acceptance, level of mindfulness, and quality of life; and
4. To study participants' characteristics related to adherence and benefits associated with MBRP.

DETAILED DESCRIPTION:
Overall Study Design This is a feasibility study and it is a single-blinded, randomized controlled trial with two study arms: the mindfulness-based relapse prevention (MBRP) programme led by trained mindfulness instructors and a usual care control group (UCCG). The MBRP will last for 8 weeks and outcome measures will be collected at similar time points in both the MBRP and UCCG groups (baseline, immediately post intervention, at 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention) . Qualitative focus group discussions or individual interviews will be conducted to obtain feedback of the MBRP programme from participants after the MBRP course. The study design, implementation and result reporting will follow the recommendations from the Standard Protocol Items Recommendations for Interventional Trials (SPIRIT), Consolidated Standards of Reporting Trials (CONSROT), and Consolidated criteria for reporting qualitative research (COREQ).

Subjects Recruitment Process To increase the representativeness of the recruited participants with substance abuse disorder, study team will recruit the study's participants from the Counselling Centres for Psychotropic Substance Abusers (CCPSAs), residential detoxification centres, other non-governmental organisations (NGOs) that provide outreach or counselling services to psychotropic substance users, and substance abuse clinics (SACs). Similar approaches for recruitment have been adopted in previous local studies. Clients who receive services at the CCPSAs or the participating NGOs and SACs will be invited to be screened by the senior research assistant (RA) to determine eligibility to enrol in the study. The senior research assistant will visit the centres to identify all eligible subjects, invite them to participate and they will then be invited to be screened further for eligibility by a clinician and obtain their written consent.

Intervention and Control Mindfulness-based Relapses Prevention (MBRP) The MBRP program will be delivered by an instructor with training in MBSR/MBCT who has more than two years of teaching experience in MBSR/MBCT. MBRP programme consists of two-and-a-half-hour weekly sessions for eight weeks with the objective and activity of each session described in Appendix A and the manualized MBRP programme will be used with each session having a central theme, with meditation practices and related relapse prevention exercises and discussions. Themes will include the concept of "automatic pilot" and its relationship to addiction relapse, recognizing thoughts and emotions in relation to triggers of relapse, integrating mindfulness practices into daily activities, practicing mindfulness skills in high risk situations and the role of thoughts and emotions in relapse. Each class will consist of between 10-12 participants. The program will also include daily homework exercises that consist of guided (taped) or unguided awareness exercises directed at increasing moment-by-moment non-judgmental awareness of bodily sensations, thoughts and feelings, together with exercises designed to integrate the application of awareness skills into daily life. The mindfulness curriculum will include training in mindfulness through (1) a body scan, the gradual moving of attention through the body from head to feet while lying on a mat on the floor, brining awareness particularly to bodily sensations; (2) sitting meditation, in which attention is brought to breathing sensations and the flow of bodily sensations, thoughts, and emotions; and (3) mindful stretching exercises, to cultivate awareness during simple stretching movement. The key themes of MBRP will include the empowerment of participants and a focus on awareness and acceptance of experience at the present moment. Participants are guided to develop a "decentered" perspective on thoughts and feelings, in which these are viewed as passing events in the mind. Two to four mindfulness instructors will be hired for the MBRP courses, which can provide with better generalisibility of the intervention.

Fidelity Check of MBRP Fidelity check will be conducted by randomly selecting 25% of the MBRP courses and scoring the courses using a checklist specifically designed for the MBRP course with reference to our previous mindfulness-based interventional course checklists.

Usual Care Control Group (UCCG) Participants in the UCCG condition will remain in their standard outpatient aftercare provided by the treatment agency with an aim to maintain their abstinence with the help from social workers or other healthcare professionals through different activities, such as topics on life training skills such as rational thinking skills, grief and loss, assertiveness, self esteem, goal setting, effects of drugs on interpersonal relationships and experience. Frequency of their visits to / contacts with healthcare professionals will be recorded.

Course Attendance, Participant Feedback and Qualitative Components Course attendances will be recorded. A questionnaire will be used to assess course satisfaction at the end of the 8 week course using a 10 point Likert scale ranging from "Not at all" to "Very". Questions will include: How important is this program to you?" and "How likely are you going to continue engaging in mindfulness practice after this course?" and "Would you recommend this course to your friends or people affected with addiction problems?". Furthermore, qualitative focus group discussions lasting for about one hour will be conducted after the course and moderated by an experienced research assistant in running focus group discussions with the support of another one in taking field notes. The discussions will be audio-recorded to ensure data accuracy. A topic guide will be used which covers open-ended questions categorized by the following topics: overall viewpoints; practice of mindfulness; perceived facilitators and barriers when applying mindfulness skills; perceived changes after the course and suggestions for improvement. For those who are not in the last course, a 30-minute individual interview through telephone will be invited. Personal preferences will be highly respected during the qualitative focus group discussions and interviews. Participants can choose to talk as much or little as they wish, or request for not recording any comments already been expressed.

All the quantitative assessments used in this study are widely used validated tools among drug users or used in our previous studies. Data will be gathered from structured interviews administered by a trained research assistant and clinician. The assessment components will include the following items.

Basic demographic data (age, sex, education, employment, marital status, district of residence, smoking and drinking status) will be collected. A trained clinician will administer the Structured Clinical Interview for DSM-5 (SCID-5 for DSM-5) to assess substance abuse and dependence and other disorders at the eligibility screening interview.

The quantitative primary and secondary outcome measures will be collected at baseline and at eight weeks (end of intervention), and at three, six, nine and twelve months after completing the MBRP by a blinded research assistant who does not know the outcome of the random group allocation.

Data analyses Descriptive statistics of the characteristics of all subjects will be computed and the demographic and clinical data of the two groups (MBRP and UCCG) will be compared via χ2 test. Student's t-tests will be employed to analyse the baseline psychological data of the two groups. Linear mixed models will be used to analyse effects of the MBRP compared to UCCG on primary and secondary outcomes, as well as potential influencing factors of the changes in outcomes, including age, sex, severity and duration of drug use, abuse of other drugs and duration of abstinence at baseline. Finally, study team will examine the correlation between the psychological parameters (secondary outcome measures) and drug craving as well as correlation between psychological parameters and drug abstinence. Intention to treat and modified intention to treat analyses would be applied. The significance level will be set at p < 0.05 (two sides).

For qualitative results, the audio recordings will be transcribed verbatim. A quality check will be completed independently by another research assistant. Framework analysis will be used by first reading through the transcripts and field notes to become familiar with the data by two researchers, then conceptualizing the themes and subthemes and piloted coding with the themes. Based on similarities and differences between initial themes, the themes and subthemes will be finalized which will include: comments on the course, home practice, changes after the course, barriers and facilitators for course participation and compliance and suggestions for course improvement. Any discrepancies will be discussed and a consensus will be reached within the team. The results will be then finally summarized and interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in Cantonese;
* Has ever fulfilled the Structured Clinical Interview for DSM-IV/DSM-5 (SCID) drug module criteria for substance use disorder diagnoses; and
* Has completed outpatient or inpatient treatment for substance abuse in the previous 6 months.

Exclusion Criteria:

* Inability to provide valid consent;
* Current or lifetime psychotic disorder assessed by the Structured Clinical interview for DSM-IV/DSM-5;
* Imminent suicidal risk; or
* Dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Self report of any drug abuse and usage | Post intervention (after 8 weeks of intervnetion from baseline)
  Self-reports of no substance use to confirm abstinence status
Urine drug test (also known as Urine drug screen or UDS) | Post intervention (after 8 weeks of intervnetion from baseline)
  Urine test for the presence of illegal drugs and prescription medications

SECONDARY OUTCOMES:
The Penn Alcohol Craving Scale | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  The Penn Alcohol Craving Scale is a 5 item, self report measure that assesses frequency, intensity and duration of craving. It has been shown to have excellent internal consistency and predictive validity for substance abuse relapse. The questions use numerical ratings from 0 to 6. Higher PACS scores represent greater craving.
the 9-item Patient Health Questionnaire (PHQ-9) | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  High reliability and validity, and widely used among different populations. The scale has four-point scales with scores ranging from 0 (rarely) to 3 (most of the time). The scores of 5 to 9, 10 to 14, 15 to 19, and 20 to 27 in PHQ-9 indicate mild, moderate, and severe depressive symptoms, respectively. A score ≥10 for the PHQ-9 indicate the presence of positive depression and anxiety symptoms, with higher scores indicating more severe symptoms.
the 7-item Generalised Anxiety Disorder (GAD-7) | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  High reliability and validity, and widely used among different populations. The scale has four-point scales with scores ranging from 0 (rarely) to 3 (most of the time). The scores of 5 to 9, 10 to 14, and 15 to 21in GAD-7 indicate mild, moderate, and severe anxiety symptoms, respectively. A score ≥10 for the GAD-7 indicate the presence of positive depression and anxiety symptoms, with higher scores indicating more severe symptoms.
The Addiction Severity Index (ASI) - Lite Version | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  A multi-dimensional interview that will be used to measure subjects' substance use, health and social problems
Drug Avoidance Self-Efficacy Scale | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  It measure self-efficacy of drug avoidance in 16 situations that may trigger someone's intention to take drugs. Responses are rated on a 7-point scale ranging from "certainly yes" to "certainly no" which corresponds to a measure of "strength" of self-efficacy. Some items are reversely coded. The total score is obtained by summing across the 16 items. Higher scores indicate higher level of self-efficacy.
The Acceptance and Action Questionnaire - second edition (AAQ-II) | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  It assesses acceptance versus avoidance and control of negative private experiences. Items of this scale are rated on a 7-point Likert-type scale, with higher scores indicating higher acceptance. Lower scores of this scale have been shown to be associated with increased levels of psychopathology and decreased quality of life.
Five Facet Mindfulness Questionnaire | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  To evaluate whether the increase or changes in mindfulness are related to changes in the outcomes
5-item EuroQol EQ-5D-5L (EQ5D) | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  Validated and widely used. It has an index score. It also has a visual analogue scale ranging from 0 to 100 with higher scores indicate better quality of life.
Meditation practice worksheet | baseline, post intervention (after 8 weeks of intervnetion from baseline), 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  Meditation practice will be recorded using a worksheet that report the type and duration of mindfulness practice to be submitted weekly to the instructors throughout and at each follow up of the study.
Self report of any drug abuse and usage | baseline, 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  Self-reports of no substance use to confirm abstinence status
Urine drug test (also known as Urine drug screen or UDS) | baseline, 3 months post intervention, 6 months post intervention, 9 months post intervention and 12 months post intervention
  Urine test for the presence of illegal drugs and prescription medications

CONTACTS AND LOCATIONS:
Overall Officials: Samuel YS Wong, Principal Investigator — JCSPHPC, CUHK
Locations (9):
- Hong Kong (9):
  - Department of Psychiatry, AHNH, Hospital Authority, Hong Kong
  - Department of Psychiatry, NDH, Hospital Authority, Hong Kong
  - Evergreen Lutheran Centre, Hong Kong Lutheran Social Service, Hong Kong
  - Neo-Health Group, Hong Kong
  - PS33 - Shamshuipo Centre, Hong Kong Christian Service, Hong Kong
  - Rainbow Lutheran Centre, Hong Kong Lutheran Social Service, Hong Kong
  - Sane Centre, Hong Kong
  - The Society of Rehabilitation and Crime Prevention, Oasis, Hong Kong
  - TWGHs CROSS Centre, Hong Kong

IPD SHARING:
Plan to Share IPD: No